CLINICAL TRIAL: NCT04152759
Title: A Randomized, Double-blinded, Single-dose, 2-arm Parallel, Comparative Study to Evaluate the Pharmacokinetics and Safety of BAT2506 Injection vs Simponi in Healthy Chinese Male Subjects
Brief Title: Comparative Study to Evaluate the Pharmacokinetics of BAT2506 vs Simponi® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-2506-001-CR
Record Dates: First submitted 2019-09-09; First posted 2019-11-05 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2019-11

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAT2506 injection (Experimental): 50mg ；subcutaneous injection
  Interventions: Drug: Drug: BAT2506 injection Other Names: Simponi(EU-licensed)
- Sinponi(EU-licensed) (Active Comparator): 50mg ；subcutaneous injection
  Interventions: Drug: Drug: BAT2506 injection Other Names: Simponi(EU-licensed)

INTERVENTIONS:
Drug: Drug: BAT2506 injection Other Names: Simponi(EU-licensed) — Drug: BAT2506 injection Each subject will receive single subcutaneous injection of 50 mg BAT2506 Injection or Simponi(EU-licensed).
  Other Names:
  Simponi(EU-licensed)
  Other Names: BAT2506

SUMMARY:
It is a randomized, double-blinded, single-dose, 2-arm parallel, comparative study to evaluate the pharmacokinetics and safety of BAT2506 Injection vs Simponi in healthy chinese male subjects A total of 182 subjects are planned to be included and randomized at a ratio of 1:1 to receive single subcutaneous administration of 50mg BAT2506 Injection or Simponi® (EU-licensed ).

The study has a screening period of 14 days. PK blood samples will be collected from subjects to determine the serum concentration of Golimumab, thus to evaluate the change and similarity of the pharmacokinetics of the two study drugs.

The investigator will perform safety evaluation for vital signs, physical examinations, injection site reaction, ECG, clinical laboratory tests and adverse events throughout the study. Immunogenicity evaluation (ADA, ADA titration and nAb) will also be evaluated.

DETAILED DESCRIPTION:
It is a randomized, double-blinded, single-dose, 2-arm parallel, comparative study to evaluate the pharmacokinetics and safety of BAT2506 Injection vs Simponi in healthy chinese male subjects A total of 182 subjects are planned to be included and randomized at a ratio of 1:1 to receive single subcutaneous administration of 50mg BAT2506 Injection or Simponi® (EU-licensed ).

The study has a screening period of 14 days. PK blood samples will be collected from subjects to determine the serum concentration of Golimumab, thus to evaluate the change and similarity of the pharmacokinetics of the two study drugs.

The investigator will perform safety evaluation for vital signs, physical examinations, injection site reaction, ECG, clinical laboratory tests and adverse events throughout the study. Immunogenicity evaluation (ADA, ADA titration and nAb) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged18 and 50 years inclusive; BMI between 18 and 28 kg/m2 and body weight between 50 and 80 kg.
* Physical examinations and vital signs are normal or abnormal without clinical significance.
* Abdominal color Doppler ultrasound, laboratory tests, etc. are normal or abnormal without clinical significance.

Exclusion Criteria:

* Any current or history of severe allergic reaction to foods or drugs and History of allergy to study products.
* Having severe injuries or surgery or fractures within 4 weeks before enrollment,or to receive surgery during the study.
* Having clinically significantclinical history abnormalities or other clinically indicated diseases (including but not limited to gastrointestinal, renal, liver, neurological, hematological, endocrine, tumor, lung, immune, mental or cardiovascular diseases).
* Having malignant tumor (excluding basal cell carcinoma who has undergone resection).
* Having clinically significant chronic or acute infections at screening/incorporation; or active infections,Includes acute and chronic infections as well as local infections (bacteria, viruses, parasites, fungi or other opportunities) Sexually infected pathogen).
* Having a history of tuberculosis or latent tuberculosis or clinical manifestations suspected of being tuberculosis(including But not limited to tuberculosis).
* Having been exposed to tuberculosis or/and suspected tuberculosis symptoms and/or signs within 3 months before screening.
* Having used simponi,or any anti-tumor necrosis factor (TNF-α) biologic preparation or any biological products within 6 months before enrollment or monoclonal antibodies within a month.
* Having used drugs within 30 days before enrollment (including but not limited to prescription drugs, Chinese medicine, non-prescription drugs).
* Having vaccinated active / attenuated vaccine within 12 weeks before screening or planned to vaccinate active /attenuated vaccine the during the study.
* Having a history of hypertension or systolic blood pressure ≥ 140 mmHg, or diastolic blood pressure ≥ at screening/inclusion90 mmHg, and it is judged abnormalities with clinical significance.
* Electrocardiogram (ECG) examination abnormalities with clinical significance;
* Having positive detection of golimumab anti-drug antibody (ADA) during screening.
* Chest orthotopic examination abnormalities with clinical significance.
* Tuberculosis enzyme-linked immunospot assay (T-SPOT. TB) positive test,
* Having any alcoholic products within 24 hours prior to the use of the study drug.
* A drug abuse test positive or a history of drug abuse over the past five years.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Endpoint：AUC0-t | 0-71days
  Pharmacokinetics Endpoint：AUC0-t
Pharmacokinetics Endpoint：Cmax | 0-71days
  Pharmacokinetics Endpoint：Cmax

SECONDARY OUTCOMES:
Pharmacokinetics Endpoint：AUC0-inf | 0-71days
  Pharmacokinetics Endpoint：AUC0-inf

CONTACTS AND LOCATIONS:
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
Only one site study

REFERENCES:
- [Derived] Wu M, Sun J, Wu D, Xu J, Wei J, Wang Z, Yu J, Li S, Zhang H, Ding Y. A Phase I, Randomized, Double-Blind, Single-Dose, Parallel-Group Study to compare Pharmacokinetic Similarity, Safety, and Immunogenicity Between BAT2506 and Golimumab in Healthy Chinese Male Subjects. Expert Opin Investig Drugs. 2021 Jan;30(1):77-83. doi: 10.1080/13543784.2021.1851364. Epub 2020 Nov 26. PMID 33241960